CLINICAL TRIAL: NCT00162864
Title: A Pilot Study of Montelukast Sodium (Singulair) in Older Adults With Asthma or Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MONTE; SING-US-75-99
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2006-03-24 (Estimated); Status verified 2005-09

CONDITIONS: Asthma; COPD
Keywords: asthma; COPD; montelukast sodium; leukotriene modifier; older adults
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — montelukast

INTERVENTIONS:
Drug: montelukast sodium

SUMMARY:
This randomized, double-blind, placebo-controlled trial assessed the efficacy of montelukast in the treatment of adults ≥50 years of age with persistent asthma and/or COPD. Primary outcomes included forced expiratory volume in one-second (FEV1) and daytime asthma symptoms scores. Nocturnal symptoms, asthma control, health-related quality of life, peak flow measurements, and health care utilization were also assessed as secondary outcomes. Participants were recruited from the Kaiser Permanente Northwest member population. One hundred forty-nine subjects were randomized to treatment with montelukast (10 mg per day) or placebo, and were followed for a six-week period. No differences in lung function measures, health-related quality of life, health care utilization, and asthma symptom scores were observed; however, the montelukast group had slightly improved asthma control scores compared to the placebo group.

DETAILED DESCRIPTION:
Asthma and COPD are common chronic conditions in older adults. Adherence to therapy is an important consideration since patients typically take two or more medications a day and often have difficulties with inhaled breathing medications. Therefore, oral preparations, such as leukotriene modifiers, have considerable appeal for older adults with asthma or COPD. Phase 3 primary studies of the leukotriene modifier, montelukast sodium (Singulair), for the management of asthma have included very few older adults.

The following randomized, double-blind, placebo-controlled study was designed as a pilot study to evaluate the efficacy of montelukast, in addition to usual therapy, in the treatment of older adults with asthma and/or COPD. Primary outcomes included pre-bronchodilator forced expiratory volume in one-second (FEV1) and average daytime asthma symptom scores.

Participants were recruited from Kaiser Permanente Northwest (KPNW), an HMO with 450,000 members in Portland, OR. All were adults ≥50 years of age with asthma and/or COPD who were symptomatic despite using daily breathing medications. They were screened by phone to collect information on asthma symptoms, medications, health care utilization, and co-morbid illnesses. Eligible persons attended a baseline visit to further assess eligibility and collect baseline data, including smoking status, co-morbidities, and participant demographics. Spirometry was performed before and twenty minutes after administration of four puffs of inhaled albuterol delivered by metered dose inhaler. All participants received instructions about the use of a peak flow meter; maintenance of a daily asthma diary with peak flow measurements, symptoms, and medications; and optimal use of an MDI by spacer.

Participants completed a two-week run-in period with placebo pills and used diaries to record peak flow each morning, use of inhaled ß-agonist, nocturnal awakenings for asthma, and occurrence of asthma attacks.

A total of 149 participants were randomized and received either montelukast(one 10 mg tablet/day) (N=71) or placebo(one tablet/day) (N=78). Spirometry was repeated at the randomization visit, and information on health status, asthma quality of life, and asthma control was collected. Participants were followed for 6 weeks after randomization. A telephone call was made at three-weeks to collect information about adverse experiences. At the final visit, participants completed spirometry, and answered questions on health status, asthma QOL and asthma control. Unscheduled health care visits for asthma during the six-week study period were noted.

Results showed that improvement in asthma control was mixed. A small improvement in the montelukast group was seen using one of the two control measures. There was no difference in lung function, asthma symptom scores, health care utilization, or health-related quality of life between the treatment and control groups.

ELIGIBILITY:
Inclusion Criteria:

* age ≥50 years
* persistent asthma symptoms
* using short-acting ß-adrenergic agonists medication
* willingness and ability to keep a daily symptom diary
* willingness to perform peak flow monitoring
* health plan membership for at least 6 months
* use of any combination of ß-agonists and inhaled corticosteroids, theophylline, cromolyn, nedocromil, or ipratropium bromide

Exclusion Criteria:

* unable to provide informed consent
* not available for duration of study
* dementia
* chronic lung disease other than asthma or COPD
* clinically significant, active disease of the gastrointestinal, cardiovascular, hepatic, neurological, renal, genitourinary, or hematologic systems
* a major surgical procedure within the four weeks prior to the baseline visit
* previous adverse reaction to montelukast
* unresolved symptoms of an upper respiratory tract infection within three weeks prior to baseline
* initiation of immunotherapy within six months before enrollment or the dose of immunotherapy was expected to change over the course of the study
* inability to adequately perform spirometry
* use of leukotriene modifiers within the past two weeks
* use of oral corticosteroids within the past 30 days
* more than one emergency department visit for asthma within the past 30 days
* more than two emergency department visits for asthma in the past six months
* hospitalization for asthma or COPD within the past six months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 1999-12; Study Completion 2002-04

PRIMARY OUTCOMES:
Forced expiratory volume in one-second (FEV1)
Daytime asthma symptoms scores

SECONDARY OUTCOMES:
Nocturnal symptoms
Asthma control
Asthma quality of life
Health status
Peak flow measurements
Health care utilization

CONTACTS AND LOCATIONS:
Overall Officials: A. Sonia Buist, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States